CLINICAL TRIAL: NCT00616590
Title: Assessment of Insomnia in Patients With Head and Neck Cancer During Treatment
Brief Title: Insomnia in Patients Undergoing Chemotherapy and Radiation Therapy for Head and Neck Cancer
Status: Withdrawn | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brittany Holmes, Medical Student, Vanderbilt University
Other Study IDs: CDR0000583565; P30CA068485 (NIH); VU-VICC-SUPP-0742
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Fatigue; Head and Neck Cancer; Psychosocial Effects of Cancer and Its Treatment; Sleep Disorders
Keywords: sleep disorders; psychosocial effects of cancer and its treatment; fatigue; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Fatigue; Head and Neck Neoplasms; Sleep Wake Disorders; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Procedure: fatigue assessment and management
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Learning about insomnia and quality of life in patients undergoing chemotherapy and radiation therapy for cancer may help doctors learn about the effects of treatment and plan the best treatment.

PURPOSE: This clinical trial is studying insomnia in patients undergoing chemotherapy and radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the prevalence of insomnia, extent of sleep disturbance, and possible contributing factors to sleep disturbance in head and neck cancer patients undergoing chemoradiotherapy.
* To evaluate the relationships between insomnia and symptom burden, quality of life, mood, fatigue, and tumor/treatment variables in these patients.

OUTLINE: Patients complete a demographic survey and a questionnaire packet comprising The Pittsburgh Sleep Quality Index, The Head and Neck Symptom Survey, Profile of Mood States, Suspected Causes of Insomnia Survey, and a Quality of Life Survey on day 1 of chemoradiotherapy to obtain baseline data on sleep quality, possible causes of sleep disruption, head and neck symptoms, mood state, fatigue, quality of life, and patient demographics. Questionnaires are administered weekly thereafter during therapy visits for up to 6-7 weeks and take 15-30 minutes to complete.

Medical records are reviewed to obtain information regarding medications and tumor- and treatment-related variables.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of head or neck carcinoma
* Currently undergoing chemoradiotherapy

PATIENT CHARACTERISTICS:

* Able to communicate in English
* Able to give informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Relationships between insomnia and symptom burden, quality of life, mood, fatigue, and tumor/treatment variables as assessed by general demographics, The Head and Neck Symptom Survey, Quality of Life Survey, and Profile of Mood States | in patient
  patient given survey while in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Holmes, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee